CLINICAL TRIAL: NCT01634763
Title: A Phase I, Multicenter, Open-label Dose Escalation Study of LDK378, Administered Orally in Japanese Patients With Tumors Characterized by Genetic Alterations in ALK
Brief Title: Study of Safety and Preliminary Efficacy for LDK378 in Japanese Patients With Genetic Alterations in Anaplastic Lymphoma Kinase (ALK)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CLDK378X1101
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-07

CONDITIONS: Tumors Characterized by Genetic Alterations in Anaplastic Lymphoma Kinase (ALK)
Keywords: Phase I, open-label, dose escalation, oral LDK378, Japanese patients with tumors characterized by ALK genetic alterations
MeSH Terms: interventions — ceritinib

ARMS (2):
- Dose-escalation (Experimental): Open-label dose escalation study of LDK378, administered orally in Japanese patients with tumors characterized by genetic alterations in anaplastic lymphoma kinase (ALK)
  Interventions: Drug: LDK378
- Dose-expansion (Experimental): Open-label study of LDK378, administered orally in Japanese patients with tumors characterized by genetic alterations in ALK to see further safety, anti-tumor activity, and PK data in patients who has progressed since prior therapy with alectinib
  Interventions: Drug: LDK378

INTERVENTIONS:
Drug: LDK378

SUMMARY:
Estimation of the Maximum tolerated dose (MTD) and/or Recommended dose (RD) of LDK378 as a single agent when administered orally to Japanese patients with tumors characterized by genetic alterations in anaplastic lymphoma kinase (ALK)

ELIGIBILITY:
Inclusion Criteria:

* Patients with a locally advanced or metastatic malignancy that has progressed despite standard therapy, or for which no effective standard therapy exists
* Only patients with tumors characterized by genetic alterations in ALK. For non-small cell lung cancer (NSCLC), an ALK translocation must be detected by Fluorescent in situ hybridization (FISH) in ≥15% of tumor cells. Local site documented results on ALK alteration are acceptable for enrollment of the patients. Central confirmation of local results is not required.

  --Eastern Cooperative Oncology Group (ECOG) performance status grade ≤ 2
* Adequate organ function
* Dose-expansion part: Patients must have NSCLC that has progressed since prior therapy with alectinib. Alectinib must have been the only prior ALK inhibitor received by the patient prior to trial entry.

Exclusion Criteria:

* Patients with symptomatic Central Nerve System (CNS) metastases who are neurologically unstable or require increasing doses of steroids to control their CNS disease
* Patients with unresolved nausea, vomiting or diarrhea > Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Other concurrent severe and/or uncontrolled medical conditions
* Patients who have been treated with chemotherapy or biologic therapy or other investigational agent < 2 weeks prior to starting the daily dosing of the study drug for compounds with a half-life ≤ 3 days, and < 4 weeks prior to starting the daily dosing of the study drug for compounds with a prolonged half-life (< 6 weeks for patients that received nitrosoureas or mitomycin-C)
* Unresolved toxicity greater than CTCAE grade 1 or unstable toxicity from previous anti-cancer therapy or radiotherapy (excluding neurotoxicity, alopecia, ototoxicity, lymphopenia), or incomplete recovery from previous surgery, unless agreed by Novartis and the Principal Investigator and documented
* Patients who have received radiotherapy to lung within 4 weeks prior to starting the daily dosing of the study drug or patients who have not recovered from radiotherapy-related toxicities. For all other anatomic sites radiotherapy to a large volume (including whole brain radiotherapy) < 2 weeks prior to starting the daily dosing of the study drug, and patients who have received radiotherapy to a small volume (including stereotactic radiotherapy to the CNS) < 3 days prior to starting the study drug.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and/or Recommended dose (RD) of LDK378 | During the first cycle (including the Pharmacokinetics [PK] run-in period) of LDK378 treatment. A treatment cycle consists of 21 days of daily dosing of LDK378.
  As a single agent when administered orally to Japanese patients with tumors characterized by genetic alterations in ALK. The number of patients and category of Dose Limiting Toxicities (DLTs)

SECONDARY OUTCOMES:
The safety and tolerability of LDK378, including both acute and chronic toxicities | Until disease progression or unacceptable toxicity occurs, or patient withdrawal
  Adverse drug reactions and serious adverse drug reactions, changes in hematology and blood chemistry values, assessments of physical examinations, vital signs and electrocardiograms
Plasma concentration of LDK378 | PK run-in (0,0.5, 1, 2, 3, 4, 6, 8, 24, 48, and 72 hrs), Cycle1Day1 (0, 0.5, 1, 2, 3, 6, 8 and 24 hrs), Cycle2Day1 (0, 1, 2, 4, 6, 8 and 24 hrs), Day1 of every subsequent cycles up to Cycle6
  Single and multiple-dose PK of LDK378
Preliminary anti-tumor activity of LDK378 | Baseline and every 6 weeks until disease progression or unacceptable toxicity occurs, or patient withdrawal
  As a single agent when administered orally to Japanese patients with tumors characterized by genetic alterations in ALK at MTD and/or RD by Computed tomography (CT) / Magnetic resonance imaging (MRI). Overall response rate (complete response [CR] or partial response [PR]) and disease control rate (CR or PR or stable disease [SD]) defined according to RECIST, duration of response and progression-free survival
PK parameter: AUClast | PK run-in (0,0.5, 1, 2, 3, 4, 6, 8, 24, 48, and 72 hrs), Cycle1Day1 (0, 0.5, 1, 2, 3, 6, 8 and 24 hrs), Cycle2Day1 (0, 1, 2, 4, 6, 8 and 24 hrs), Day1 of every subsequent cycles up to Cycle6
  Single and multiple-dose PK of LDK378
PK parameter: AUCtau | PK run-in (0,0.5, 1, 2, 3, 4, 6, 8, 24, 48, and 72 hrs), Cycle1Day1 (0, 0.5, 1, 2, 3, 6, 8 and 24 hrs), Cycle2Day1 (0, 1, 2, 4, 6, 8 and 24 hrs), Day1 of every subsequent cycles up to Cycle6
  Single and multiple-dose PK of LDK378
PK parameter: Cmax | PK run-in (0,0.5, 1, 2, 3, 4, 6, 8, 24, 48, and 72 hrs), Cycle1Day1 (0, 0.5, 1, 2, 3, 6, 8 and 24 hrs), Cycle2Day1 (0, 1, 2, 4, 6, 8 and 24 hrs), Day1 of every subsequent cycles up to Cycle6
  Single and multiple-dose PK of LDK378
PK parameter: Tmax | PK run-in (0,0.5, 1, 2, 3, 4, 6, 8, 24, 48, and 72 hrs), Cycle1Day1 (0, 0.5, 1, 2, 3, 6, 8 and 24 hrs), Cycle2Day1 (0, 1, 2, 4, 6, 8 and 24 hrs), Day1 of every subsequent cycles up to Cycle6
  Single and multiple-dose PK of LDK378
PK parameter: the apparent elimination half-life (T1/2) | PK run-in (0,0.5, 1, 2, 3, 4, 6, 8, 24, 48, and 72 hrs), Cycle1Day1 (0, 0.5, 1, 2, 3, 6, 8 and 24 hrs), Cycle2Day1 (0, 1, 2, 4, 6, 8 and 24 hrs), Day1 of every subsequent cycles up to Cycle6
  Single and multiple-dose PK of LDK378
PK parameter: accumulation ratio (Racc) | PK run-in (0,0.5, 1, 2, 3, 4, 6, 8, 24, 48, and 72 hrs), Cycle1Day1 (0, 0.5, 1, 2, 3, 6, 8 and 24 hrs), Cycle2Day1 (0, 1, 2, 4, 6, 8 and 24 hrs), Day1 of every subsequent cycles up to Cycle6
  Single and multiple-dose PK of LDK378

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Japan (3):
  - Novartis Investigative Site, Sunto-gun, Shizuoka
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Fukuoka

REFERENCES:
- [Derived] Ono A, Murakami H, Serizawa M, Wakuda K, Kenmotsu H, Naito T, Taira T, Koh Y, Ohde Y, Nakajima T, Endo M, Takahashi T. Drastic initial response and subsequent response to two ALK inhibitors in a patient with a highly aggressive ALK-rearranged inflammatory myofibroblastic tumor arising in the pleural cavity. Lung Cancer. 2016 Sep;99:151-4. doi: 10.1016/j.lungcan.2016.07.002. Epub 2016 Jul 5. PMID 27565932
- [Derived] Nishio M, Murakami H, Horiike A, Takahashi T, Hirai F, Suenaga N, Tajima T, Tokushige K, Ishii M, Boral A, Robson M, Seto T. Phase I Study of Ceritinib (LDK378) in Japanese Patients with Advanced, Anaplastic Lymphoma Kinase-Rearranged Non-Small-Cell Lung Cancer or Other Tumors. J Thorac Oncol. 2015 Jul;10(7):1058-66. doi: 10.1097/JTO.0000000000000566. PMID 26020125
- See also: Results for CLDK378X1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=15487